CLINICAL TRIAL: NCT04227054
Title: Abdominal Aortic Aneurysm Sac Healing and Prevention of Endoleaks - A Prospective Single Center Safety Study
Brief Title: Abdominal Aortic Aneurysm Sac Healing and Prevention of Endoleaks
Acronym: AAA-SHAPE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shape Memory Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRD1015
Record Dates: First submitted 2020-01-10; First posted 2020-01-13 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Intervention (Experimental)
  Interventions: Device: IMPEDE-FX Embolization Plug

INTERVENTIONS:
Device: IMPEDE-FX Embolization Plug — Fill an abdominal aortic aneurysm (AAA) sac outside of an endovascular aneurysm repair (EVAR) stent graft

SUMMARY:
To determine the safety and efficacy of IMPEDE-FX Embolization Plug and/or IMPEDE-FX Rapid Fill to fill an abdominal aortic aneurysm (AAA) sac outside of an endovascular aneurysm repair (EVAR) stent graft.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* A candidate for elective EVAR of an infrarenal aortic aneurysm ≥5.5 cm in diameter in men and ≥5.0 cm in women

Exclusion Criteria:

* An inability to provide informed consent
* Enrolled in another clinical study
* Concomitant iliac artery ectasia or aneurysm (common iliac artery diameter >24 mm)
* Patent AAA sac feeding vessels (within the sac) >4 mm in diameter
* Volume of AAA sac to be filled after stent graft placement <30 mL or >135 mL, based on pre-procedure CTA (i.e. aortic flow volume exclusive of stent graft volume)
* Use of aortic stent grafts other than the Gore Excluder AAA Endoprosthesis, Cook Zenith Flex AAA Endovascular Graft, Medtronic Endurant II Stent Graft, or Endologix Ovation Alto Abdominal Stent Graft System to treat the AAA
* Planned use of the chosen stent graft outside its instructions for use (IFU)
* Planned use of fenestrated or chimney stent grafts
* Study participants in which stent graft placement is abandoned for any reason, and/or in which the investigator decides, during the course of the stent graft placement, that the study procedure may not be appropriate
* Planned use of embolic devices other than the investigational product to embolize the AAA sac
* Vascular disease and/or anatomy that preclude the safe access and positioning of a catheter to deliver the investigational product into the AAA sac
* Ruptured, leaking, or mycotic (infected) aneurysm
* Aneurysmal disease of the descending thoracic aorta
* Coagulopathy or uncontrolled bleeding disorder
* Long-term (>6 months prior to the procedure) use of direct oral anticoagulant or any vitamin K antagonist anticoagulant use
* Serum creatinine level >2.5 mg/dL;
* Cerebrovascular accident within 3 months prior to the procedure
* Myocardial infarction and/or major heart surgery within 3 months prior to the procedure
* Atrial fibrillation that is not well rate controlled
* Unable or unwilling to comply with study follow-up requirements
* Life expectancy of <2 years post-procedure
* Known hypersensitivity or contraindication to platinum, iridium, or polyurethane
* A condition that inhibits radiographic visualization during the implantation procedure
* History of allergy to contrast medium that cannot be managed medically
* Uncontrolled co-morbid medical condition, including mental health issues, that would adversely affect participation in the study
* Pregnant or a lactating female. For females of child-bearing potential, based on a positive pregnancy test within 7 days prior to the procedure or refusal to use a medically accepted method of birth control for the duration of the study
* Prisoner or member of other vulnerable population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-09-09 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of related major adverse events (MAEs) | 30 days post-procedure
  Incidence of related major adverse events (MAEs)
Efficacy - Technical Success | Immediately after the intervention
  Technical success, defined as filling of the residual flow lumen of the AAA sac with investigational products

SECONDARY OUTCOMES:
Incidence of related major adverse events (MAEs) | 5 years post-procedure
  Incidence of related major adverse events (MAEs)
Incidence of related serious adverse events (SAEs) | 5 years post-procedure
  Incidence of related serious adverse events (SAEs)
Efficacy - Type II endoleaks | 5 years post-procedure
  Incidence of type II endoleaks
Efficacy - Type I and type III endoleaks | 5 years post-procedure
  Incidence of type I and type III endoleaks
Efficacy - AAA sac diameter/volume | 5 years post-procedure
  Change in AAA sac diameter/volume
Efficacy - Open repair | 5 years post-procedure
  Rate of conversion to open AAA repair
Efficacy - Reinterventions | 5 years post-procedure
  Rate of other reinterventions related to the AAA sac growth and/or complications

CONTACTS AND LOCATIONS:
Locations (2):
- New Zealand (2):
  - Auckland City Hospital, Auckland, Auckland
  - Waikato Hospital, Hamilton

IPD SHARING:
Plan to Share IPD: No